CLINICAL TRIAL: NCT03698994
Title: NCI-COG Pediatric MATCH (Molecular Analysis for Therapy Choice) - Phase 2 Subprotocol of BVD-523FB (Ulixertinib) in Patients With Tumors Harboring Activating MAPK Pathway Mutations
Brief Title: Ulixertinib in Treating Patients With Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Histiocytic Disorders With MAPK Pathway Mutations (A Pediatric MATCH Treatment Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02150; NCI-2018-02150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APEC1621J (Other: Children's Oncology Group); APEC1621J (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Recurrent Ependymal Tumor; Recurrent Ewing Sarcoma; Recurrent Glioma; Recurrent Hepatoblastoma; Recurrent Histiocytic and Dendritic Cell Neoplasm; Recurrent Langerhans Cell Histiocytosis; Recurrent Malignant Germ Cell Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Peripheral Primitive Neuroectodermal Tumor; Recurrent Primary Malignant Central Nervous System Neoplasm; Recurrent Rhabdoid Tumor; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Refractory Ependymoma; Refractory Ewing Sarcoma; Refractory Glioma; Refractory Hepatoblastoma; Refractory Histiocytic and Dendritic Cell Neoplasm; Refractory Langerhans Cell Histiocytosis; Refractory Malignant Germ Cell Tumor; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Peripheral Primitive Neuroectodermal Tumor; Refractory Primary Malignant Central Nervous System Neoplasm; Refractory Rhabdoid Tumor; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Wilms Tumor
MeSH Terms: conditions — Sarcoma, Ewing; Glioma; Hepatoblastoma; Histiocytosis, Langerhans-Cell; Medulloblastoma; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Rhabdoid Tumor; Rhabdomyosarcoma; Sarcoma; Ependymoma; Wilms Tumor | interventions — Pharmacogenomic Variants; ulixertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ulixertinib) (Experimental): Patients receive ulixertinib PO BID. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Pharmacokinetic Study; Drug: Ulixertinib

INTERVENTIONS:
Other: Pharmacokinetic Study — Ancillary studies
  Other Names: PHARMACOKINETIC; PK Study
Drug: Ulixertinib — Given PO
  Other Names: BVD-523; VRT752271

SUMMARY:
This phase II Pediatric MATCH trial studies how well ulixertinib works in treating patients with solid tumors that have spread to other places in the body (advanced), non-Hodgkin lymphoma, or histiocytic disorders that have a genetic alteration (mutation) in a signaling pathway called MAPK. A signaling pathway consists of a group of molecules in a cell that control one or more cell functions. Genes in the MAPK pathway are frequently mutated in many types of cancers. Ulixertinib may stop the growth of cancer cells that have mutations in the MAPK pathway.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate (ORR; complete response + partial response) in pediatric patients treated with BVD-523FB (ulixertinib) with advanced solid tumors (including central nervous system [CNS] tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor activating genetic alterations in the MAPK pathway.

SECONDARY OBJECTIVES:

I. To estimate the progression free survival in pediatric patients treated with BVD-523FB (ulixertinib) with advanced solid tumors (including CNS tumors), non-Hodgkin lymphomas or histiocytic disorders that harbor activating genetic alterations in the MAPK pathway.

II. To obtain information about the tolerability of BVD-523FB (ulixertinib) in children and adolescents with relapsed or refractory cancer.

III. To provide preliminary estimates of the pharmacokinetics of BVD-523FB (ulixertinib) in children and adolescents with relapsed or refractory cancer.

EXPLORATORY OBJECTIVES:

I. To evaluate other biomarkers as predictors of response to BVD-523FB (ulixertinib) and specifically, whether tumors that harbor different mutations or fusions will demonstrate differential response to BVD-523FB (ulixertinib) treatment.

II. To explore approaches to profiling changes in tumor genomics over time through evaluation of circulating tumor deoxyribonucleic acid (DNA).

OUTLINE: This is a dose-escalation study.

Patients receive ulixertinib orally (PO) twice daily (BID). Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto APEC1621SC and must have been given a treatment assignment to MATCH to APEC1621J based on the presence of an actionable mutation.
* Patients must have a body surface area >= 0.54 m^2 at the time of study enrollment.
* Patients must have radiographically measurable disease at the time of study enrollment. Patients with neuroblastoma who do not have measurable disease but have metaiodobenzylguanidine (MIBG)+ evaluable disease are eligible. Measurable disease in patients with central nervous system (CNS) involvement is defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI) and visible on more than one slice.

  * Note: The following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by MIBG scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted for neuroblastoma
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement requirements for Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately.

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive.

    * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or ANC counts): >= 7 days after the last dose of agent.
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1.
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid.
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For growth factors that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair and the study-assigned research coordinator.
  * Interleukins, Interferons and Cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors).
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including DLI or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD).
    * Autologous stem cell infusion including boost infusion: >= 42 days.
  * Cellular Therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.).
  * Radiotherapy (XRT)/External Beam Irradiation including Protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial brain metastases (BM) radiation.

    * Note: Radiation may not be delivered to "measurable disease" tumor site(s) being used to follow response to subprotocol treatment.
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days after systemically administered radiopharmaceutical therapy.
  * Patients must not have received prior exposure to BVD-523FB (ulixertinib) or other ERK inhibitors.
* For patients with solid tumors without known bone marrow involvement: Peripheral absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days prior to enrollment).
* For patients with solid tumors without known bone marrow involvement: Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions). These patients will not be evaluable for hematologic toxicity.
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2, or (within 7 days prior to enrollment).
* A serum creatinine based on age/gender (within 7 days prior to enrollment).

  * Age 1 to < 2 years, maximum serum creatinine (mg/dL) male 0.6, female 0.6
  * Age 2 to < 6 years, maximum serum creatinine (mg/dL) male 0.8, female 0.8
  * Age 6 to < 10 years, maximum serum creatinine (mg/dL) male 1, female 1
  * Age 10 to < 13 years, maximum serum creatinine (mg/dL) male 1.2, female 1.2
  * Age 13 to < 16 years, maximum serum creatinine (mg/dL) male 1.5, female 1.4
  * Age >= 16 years, maximum serum creatinine (mg/dL) male 1.7, female 1.4
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment).
* Serum glutamate-pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L. (For the purpose of this study, the ULN for SGPT is 45 U/L.) (within 7 days prior to enrollment).
* Serum albumin >= 2 g/dL (within 7 days prior to enrollment).
* Shortening fraction of >= 27% by echocardiogram, or (within 7 days prior to enrollment).
* Ejection fraction of >= 50% by gated radionuclide study (within 7 days prior to enrollment).
* QTc interval =< 480 milliseconds (within 7 days prior to enrollment).
* Patients must be able to swallow intact capsules.
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study treatment and for 3 months after last dose of BVD-523FB (ulixertinib).
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid.
* Patients who are currently receiving another investigational drug are not eligible.
* Patients who are currently receiving other anti-cancer agents are not eligible.
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial.
* Patients who are currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided from 14 days prior to enrollment to the end of the study. Note: CYP3A4 inducing anti-epileptic drugs and dexamethasone for CNS tumors or metastases, on a stable dose, are allowed.
* Patients who are currently receiving drugs that are strong inducers or inhibitors of CYP1A2 and CYP2D6 are not eligible. Strong inhibitors of CYP1A2 (e.g., ciprofloxacin, enoxacin, fluvoxamine, zafirlukast) should be avoided from 14 days prior to enrollment to the end of the study. Strong inhibitors of CYP2D6 (e.g., bupropion, paroxetine, fluoxetine, quinidine, terbinafine) should also be avoided from 14 days prior to enrollment to the end of the study.
* Patients with known significant ophthalmologic conditions (uncontrolled glaucoma, history of retinal vein occlusion or retinal detachment, excluding patients with longstanding findings secondary to existing conditions) are not eligible.
* Patients who have an uncontrolled infection are not eligible.
* Patients who have received a prior solid organ transplantation are not eligible.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kieuhoa T Vo, Principal Investigator — Children's Oncology Group
Locations (107):
- United States (105):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ulixertinib)
Started | 20
Completed | 1
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ulixertinib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR = Complete Response [CR] + Partial Response [PR]) in Pediatric Patients Treated With BVD-523FB (Ulixertinib)
Description: ORR will be defined as complete response + partial response and assessed by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Response rates will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed using the Wilson score interval method.
Time Frame: From enrollment to the end of treatment, up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ulixertinib)
Number analyzed (Participants) | 20
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Progression Free Survival (PFS) in Pediatric Patients Treated With Ulixertinib
Description: PFS along with the confidence intervals will be estimated using the Kaplan-Meier method.
Time Frame: From initiation of treatment to disease progression, disease recurrence, or death from any cause assessed up to 2 years
Reporting Status: Not Posted, anticipated posting 2027-01

3. Secondary Outcome: Percentage of Patients Experiencing Grade 3 or 4 Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Any eligible patient who receives at least one dose of protocol therapy will be considered in the evaluation of toxicity.
Time Frame: From enrollment to the end of treatment, up to 2 years
Reporting Status: Not Posted, anticipated posting 2027-01

4. Secondary Outcome: Preliminary Estimates of the Pharmacokinetics of Ulixertinib in Children and Adolescents With Relapsed or Refractory Cancer
Description: Will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Time Frame: Pre-dose and 1, 2, 4, and 6-8 hours after dose on cycle 1, day 1; and pre-dose on cycle 1, day 2, and cycle 1, day 15
Reporting Status: Not Posted, anticipated posting 2027-01

5. Other Pre Specified Outcome: Other Biomarkers as Predictors of Response to Ulixertinib and Whether Tumors That Harbor Different Mutations or Fusions Will Demonstrate Differential Response to Treatment
Description: Will be performed and will be summarized with simple summary statistics. All of these analyses will be descriptive in nature.
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Profiling Changes in Tumor Genomics Over Time Through Evaluation of Circulating Tumor Deoxyribonucleic Acid (DNA)
Description: as for outcome 5
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From enrollment to 30 days after the end of treatment, up to 2 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Treatment (Ulixertinib)
All-Cause Mortality (participants affected / at risk) | 4/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ulixertinib) (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ulixertinib) (N=20)
Anemia (Blood and lymphatic system disorders) | 11
Eosinophilia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 4
Blurred vision (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 5
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 1
Edema face (General disorders) | 2
Edema limbs (General disorders) | 2
Facial pain (General disorders) | 1
Fatigue (General disorders) | 9
Fever (General disorders) | 7
Generalized edema (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Eye infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 11
Blood bicarbonate decreased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 6
Ejection fraction decreased (Investigations) | 1
INR increased (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 4
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 6
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Superficial thrombophlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03698994/Prot_SAP_000.pdf